CLINICAL TRIAL: NCT05475535
Title: Can a Self-guided Cognitive Behavioral-based Mobile Phone Application Program With a Self-Compassion Component Reduce Unhealthy Perfectionism in University Students - a Randomised Controlled Trial (RCT) With a 4-week Follow-up
Brief Title: Can a Self-guided Mobile Phone Application Program Improve Wellbeing in University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Tan Pei En Marie, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NUS-IRB-2022-307
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Perfectionism; Shame; Depression, Anxiety; Stress; Self-Compassion
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Control (Active Comparator)
  Interventions: Behavioral: Active Control
- Cognitive Behavioural Therapy (CBT) (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Self-Compassion (SC) (Experimental)
  Interventions: Behavioral: Self-Compassion
- Cognitive Behavioural Therapy and Self-Compassion (CBT+SC) (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Therapy; Behavioral: Self-Compassion

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Cognitive Behavioural Therapy
  Arms: Cognitive Behavioural Therapy (CBT); Cognitive Behavioural Therapy and Self-Compassion (CBT+SC)
Behavioral: Self-Compassion — Self-Compassion focused exercises
  Arms: Cognitive Behavioural Therapy and Self-Compassion (CBT+SC); Self-Compassion (SC)
Behavioral: Active Control — Engagement in a mobile application (Cooperation skills)
  Arms: Active Control

SUMMARY:
This study seeks to evaluate and compare the effectiveness of a mobile phone application-based intervention in improving wellbeing in young adults. 400 University students are randomized into 1 of 4 intervention types. Pre, mid and post-intervention outcome measures are compared to determine effectiveness of the various intervention types.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone with the following requirements: iPhone 8 and above, or Android 5.2+ (display greater than 5 inches)
* Have scores of greater than or equal to 29 on the 'Concerns over Mistakes' subscale on the FMPS

Exclusion Criteria:

* Participants who do not meet the inclusion criteria
* Currently pregnant
* Undergoing psychological treatment or counselling
* Have any change in psychotropic medication within twelve weeks before starting intervention

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in maladaptive perfectionism | Day 1, Day 8, Day 14, 4 weeks after completion of treatment
  Frost Multidimensional Perfectionism Scale (FMPS). A 35-item self-report questionnaire which assesses four sub-scales of perfectionism - Concern over mistakes, Excessive concern with parental expectations, Personal Standards and Concern with precision, order and organisation. It is scored on a five-point scale, from "Strongly disagree" (1) to "Strongly agree" (5). Higher scores reflect higher levels of maladaptive perfectionism.
Change in shame | Day 1, Day 8, Day 14, 4 weeks after completion of treatment
  Internalized Shame Scale (ISS). A 30-item self-report questionnaire which assesses internalized shame, and a subscale of self-esteem. It is scored on a five-point scale from "Never" (1) to "Almost always" (5). Higher scores reflect greater symptom severity.
Change in Self-Compassion | Day 1, Day 8, Day 14, 4 weeks after completion of treatment
  Self-Compassion Scale (SCS-SF). A 12-item self-report questionnaire which assesses degree of self-compassion. It is the briefer version of the Self-Compassion Scale (SCS) (Neff, 2003). It is scored on a five-point scale from "Almost never" (1) to "Almost all of the time" (5). A total score is derived from taking the mean of the 12 items. Higher scores reflect greater self- compassion.

SECONDARY OUTCOMES:
Change in Depression | Day 1, Day 8, Day 14, 4 weeks after completion of treatment
  Depression, Anxiety, Stress Scale - 21 (DASS-21). A 21-item self-report questionnaire, which comprises of 3 subscales which assess levels of depression, anxiety and stress. It is scored on a four-point scale, from "Did not apply to me at all" (0) to "Applied to me very much or most of the time" (3). Higher scores reflect greater symptom severity.
Change in Anxiety | Day 1, Day 8, Day 14, 4 weeks after completion of treatment
  Depression, Anxiety, Stress Scale - 21 (DASS-21). A 21-item self-report questionnaire, which comprises of 3 subscales which assess levels of depression, anxiety and stress. It is scored on a four-point scale, from "Did not apply to me at all" (0) to "Applied to me very much or most of the time" (3). Higher scores reflect greater symptom severity.
Change in Stress | Day 1, Day 8, Day 14, 4 weeks after completion of treatment
  Depression, Anxiety, Stress Scale - 21 (DASS-21). A 21-item self-report questionnaire, which comprises of 3 subscales which assess levels of depression, anxiety and stress. It is scored on a four-point scale, from "Did not apply to me at all" (0) to "Applied to me very much or most of the time" (3). Higher scores reflect greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Tan, Principal Investigator — National University of Singapore

IPD SHARING:
Plan to Share IPD: No